CLINICAL TRIAL: NCT03780543
Title: A Multi-center, Open-label, Long-term Extension Study of ABI-H0731 + Nucleos(t)Ide as Finite Treatment for Chronic Hepatitis B Patients
Brief Title: A Study of ABI-H0731 + Nucleos(t)Ide as Finite Treatment for Chronic Hepatitis B Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-H0731-211; NCT03780543 (Registry Identifier: ClinicalTrials.gov identifier)
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-02

CONDITIONS: Chronic Hepatitis B
Keywords: CHB (chronic hepatitis B infection); HBV (hepatitis B virus); HBeAg positive (hepatitis B "e" antigen - positive); HBeAg negative (hepatitis B "e" antigen - negative); Hepatitis B (hepatitis B virus); Hepatitis B virus (HBV); SVR (sustained viral response)
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Standard of Care; entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HBeAg-negative Subjects from Parent Study ABI-H0731-201 (Active Comparator): Subjects who on Day 1 of parent study ABI-H0731-201 (NCT03576066) were standard of care (SOC) nucleos(t)ide (NrtI)-suppressed and HBeAg-negative will receive both ABI-H0731 + SOC NrtI for at least 52 weeks, after which time they will discontinue both ABI-H0731 and SOC NrtI and enter long-term off-treatment follow-up (FU) for up to 3 years.
  Interventions: Drug: standard of care (SOC) Nucleoside reverse transcriptase inhibitor (NrtI)
- HBeAg-positive Subjects from Parent Study ABI-H0731-201 (Active Comparator): Subjects who on Day 1 of parent study ABI-H0731-201 (NCT03576066) were SOC NrtI-suppressed and HBeAg-positive will receive ABI-H0731 + SOC NrtI for at least 52 weeks, after which time their viral response will be evaluated.
  1. Subjects who meet the virologic response criteria will discontinue both ABI-H0731 and SOC NrtI and enter long-term off-treatment follow-up (FU) for up to 3 years.
  2. Subjects with insufficient virologic response will discontinue ABI-H0731 only and continue on SOC NrtI alone and followed-up for 12 weeks.
  Interventions: Drug: standard of care (SOC) Nucleoside reverse transcriptase inhibitor (NrtI)
- Subjects from Parent Study ABI-H0731-202 (Active Comparator): Subjects who on Day 1 of parent study ABI-H0731-202 (NCT03577171) were treatment-naive and HBeAg-positive will receive ABI-H0731 + SOC NrtI for at least 52 weeks, after which time their viral response will be evaluated.
  1. Subjects who meet the virologic response criteria at Week 52 will continue to receive ABI-H0731 + SOC NrtI for an additional 96 weeks, after which time their viral response will be evaluated at Week 148.
     Subjects who meet the virologic response criteria at Week 148 will discontinue both ABI-H0731 and SOC NrtI and enter long-term off-treatment follow-up for up to 3 years. Subjects with insufficient virologic response at Week 148, will discontinue ABI-H0731 only and continue on SOC NrtI alone for up to 12 weeks.
  2. Subjects with insufficient virologic response at Week 52 will discontinue from ABI-H0731only and continue on SOC NrtI alone and enter follow-up for up to 12 weeks.
  Interventions: Drug: standard of care (SOC) Nucleoside reverse transcriptase inhibitor (NrtI)

INTERVENTIONS:
Drug: standard of care (SOC) Nucleoside reverse transcriptase inhibitor (NrtI) — Participants will continue on their SOC NrtI, Entecavir (ETV), Tenofovir Disoproxil Fumarate (TDF) or Tenofovir Alafenamide (TAF) tablet QD (once daily) orally as per approved package insert.
  Other Names: Entecavir (ETV) - brand name Baraclude; Tenofovir Disoproxil Fumarate (TDF) - brand name: Viread; Tenofovir Alafenamide (TAF) - brand name: Descovy

SUMMARY:
Open-label, extension study to evaluate the safety and efficacy of combination therapy and its effect on sustained viral response biomarkers.

DETAILED DESCRIPTION:
This is an open-label extension of parent studies ABI-H0731-201 (NCT03576066) and ABI-H0731-202 (NCT03577171). The extension study will assess the safety of long-term (up to 100 weeks of treatment in extension study ABI-H0731-211) combination therapy and its effect on biomarkers of sustained viral response (SVR) (NCT03780543).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. Previously enrolled on Study ABI-H0731-201 (NCT03576066) or ABI-H0731-202 (NCT03577171) and completed the treatment period, with demonstrated compliance in the opinion of the investigator.
3. Female subjects must agree to use an effective birth control method for the duration of the study and follow-up, or be surgically sterile for at least 6 months, or at least 2 years postmenopausal with serum follicle-stimulating hormone (FSH) levels consistent with a postmenopausal status. Effective birth control methods include male or female condom (may not be used together due to increased risk of breakage), vasectomy, intrauterine device (IUD), diaphragm, or cervical cap. Female subjects of childbearing potential must have a negative serum pregnancy test.
4. All heterosexually active male subjects must agree to use an effective birth control method for the duration of the study and follow-up. Effective birth control methods include male or female condom (may not be used together due to increased risk of breakage), vasectomy, hormone-based contraception (only female partner of a male subject), IUD, diaphragm, or cervical cap.
5. Agreement to adhere to Lifestyle Considerations (including abstaining from alcohol abuse [defined as alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol)] and the use of illicit substances, herbal or other substances, or unnecessary over-the-counter medications throughout study duration.
6. In good general health except for chronic HBV infection.
7. Have the ability to take oral medication and be willing to adhere to the ABI-H0731-211 regimen in the opinion of the Investigator.

Exclusion Criteria:

1. Must not have had evidence of HBV resistance-associated variants (RAVs) or lack of compliance on a previous study of ABI H0731.
2. Must not have had a treatment-emergent adverse event or laboratory abnormalities deemed clinically significant and possibly or probably related to drug while on a previous study of ABI-H0731, that in the opinion of the Investigator or the Sponsor makes the subject unsuitable for this study.
3. Current clinically significant cardiac or pulmonary disease, chronic or recurrent renal or urinary tract disease, liver disease other than HBV, endocrine disorder, autoimmune disorder, diabetes mellitus requiring treatment with insulin or hypoglycemic agents, neuromuscular, musculoskeletal, or mucocutaneous conditions requiring frequent treatment, seizure disorders requiring treatment, or other medical conditions requiring frequent medical management or pharmacologic or surgical treatment that in the opinion of the Investigator or the Sponsor makes the subject unsuitable for the study.
4. Females who are lactating or pregnant or wish to become pregnant within the duration of the ABI-H0731-211 study.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Anderson, Study Director — Assembly Biosciences Inc.; M. F. Yuen, MD, PhD, DSc, Study Chair — The University of Hong Kong
Locations (24):
- United States (17):
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - Southern California Research Center, Coronado, California
  - Coalition of Inclusive Medicine, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Research and Education, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Miami Hospital and Clinics, Miami, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Digestive Disease Associates, Catonsville, Maryland
  - Infectious Disease Care, Hillsborough, New Jersey
  - Sing Chan, MD, Flushing, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Xiaoli Ma, MD, Philadelphia, Pennsylvania
- Canada (3):
  - GI Research Institute, Vancouver, British Columbia
  - Toronto Liver Center, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong
- New Zealand (2):
  - Auckland Clinical Studies, Auckland
  - Waikato Hospital, Hamilton
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuen MF, Fung S, Ma X, Nguyen TT, Hassanein T, Hann HW, Elkhashab M, Nahass RG, Park JS, Jacobson IM, Ayoub WS, Han SH, Gane EJ, Zomorodi K, Yan R, Ma J, Knox SJ, Stamm LM, Bonacini M, Weilert F, Ramji A, Bennett M, Ravendhran N, Chan S, Dieterich DT, Kwo PY, Schiff ER, Bae HS, Lalezari J, Agarwal K, Sulkowski MS. Long-term open-label vebicorvir for chronic HBV infection: Safety and off-treatment responses. JHEP Rep. 2024 Jan 18;6(4):100999. doi: 10.1016/j.jhepr.2023.100999. eCollection 2024 Apr. PMID 38510983

RESULTS

PARTICIPANT FLOW:
Groups:
- Virologically Suppressed HBeAg-negative Participants From Parent Study ABI-H0731-201: Subjects who on Day 1 of parent study ABI-H0731-201 (NCT03576066) were standard of care nucleos(t)ide (SOC NrtI)-suppressed and HBeAg-negative will receive ABI-H0731 + SOC NrtI for at least 52 weeks, after which time they will discontinue both ABI-H0731 and SOC NrtI and be monitored for up to 3 years.
  ABI-H0731: Participants will receive 300 mg quaque die (QD) of ABI-H0731 tablets orally.
  SOC NrtI: Participants will continue on their SOC NrtI (ETV, TDF or TAF) tablet QD orally as per approved package insert.
- Virologically Suppressed HBeAg-positive Participants From Parent Study ABI-H0731-201: Subjects who on Day 1 of parent study ABI-H0731-201 (NCT03576066) were SOC NrtI-suppressed and HBeAg-positive will receive ABI-H0731 + SOC NrtI for at least 52 weeks, after which time their viral response will be evaluated. Subjects who meet the virologic response criteria will discontinue both ABI-H0731 and SOC NrtI and be monitored for up to 3 years. Subjects with insufficient virologic response will discontinue from ABI-H0731 and continue on SOC NrtI for 12 weeks.
  ABI-H0731: Participants will receive 300 mg QD of ABI-H0731 tablets orally.
  SOC NrtI: Participants will continue on their SOC NrtI (ETV, TDF or TAF) tablet QD orally as per approved package insert.
- HBeAg Positive Participants From Parent Study ABI-H0731-202: Subjects who on Day 1 of parent study ABI-H0731-202 (NCT03577171) were treatment-naive and HBeAg-positive will receive ABI-H0731 + SOC NrtI for at least 52 weeks, after which time their viral response will be evaluated.
  Subjects who meet the virologic response criteria at Week 52 will continue to receive ABI-H0731 + SOC NrtI for an additional 96 weeks, after which time their viral response will be evaluated at Week 148. Subjects who meet the virologic response criteria at Week 148 will discontinue both ABI-H0731 and SOC NrtI and be monitored for up to 3 years, while those subjects with insufficient virologic response will discontinue from ABI-H0731 and continue on SOC NrtI for 12 weeks.
  Subjects with insufficient virologic response at Week 52 will discontinue from ABI-H0731 and continue on SOC NrtI for 12 weeks.
  ABI-H0731: Participants will receive 300 mg quaque die (QD) of ABI-H0731 tablets orally.
  SOC NrtI: Participants will continue on their SOC NrtI (Entecavir (ETV), Tenofovir Disoproxil Fumarate (TDF) or Tenofovir alafenamide (TAF) tablet QD orally as per approved package insert.
Period: Overall Study
Arm/Group | Virologically Suppressed HBeAg-negative Participants From Parent Study ABI-H0731-201 | Virologically Suppressed HBeAg-positive Participants From Parent Study ABI-H0731-201 | HBeAg Positive Participants From Parent Study ABI-H0731-202
Started | 26 | 43 | 23
Completed | 13 | 28 | 6
Not Completed | 13 | 15 | 17
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Study terminated by Sponsor | 8 | 7 | 13
Not completed — Withdrawal by Subject | 1 | 8 | 1
Not completed — Noncompliance with study drug | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Virologically Suppressed HBeAg-negative Participants From Parent Study ABI-H0731-201: Subjects who on Day 1 of parent study ABI-H0731-201 (NCT03576066) were standard of care nucleos(t)ide (SOC NrtI)-suppressed and HBeAg-negative will receive ABI-H0731 + SOC NrtI for at least 52 weeks, after which time they will discontinue both ABI-H0731 and SOC NrtI and be monitored for up to 3 years.
  ABI-H0731: Participants will receive 300 mg QD of ABI-H0731 tablets orally.
  SOC NrtI: Participants will continue on their SOC NrtI (ETV, TDF or TAF) tablet QD orally as per approved package insert.
- HBeAg Positive Participants From Parent Study ABI-H0731-202: Subjects who on Day 1 of parent study ABI-H0731-202 (NCT03577171) were treatment-naive and HBeAg-positive will receive ABI-H0731 + SOC NrtI for at least 52 weeks, after which time their viral response will be evaluated.
  Subjects who meet the virologic response criteria at Week 52 will continue to receive ABI-H0731 + SOC NrtI for an additional 96 weeks, after which time their viral response will be evaluated at Week 148. Subjects who meet the virologic response criteria at Week 148 will discontinue both ABI-H0731 and SOC NrtI and be monitored for up to 3 years, while those subjects with insufficient virologic response will discontinue from ABI-H0731 and continue on SOC NrtI for 12 weeks.
  Subjects with insufficient virologic response at Week 52 will discontinue from ABI-H0731 and continue on SOC NrtI for 12 weeks.
  ABI-H0731: Participants will receive 300 mg QD of ABI-H0731 tablets orally.
  SOC NrtI: Participants will continue on their SOC NrtI (ETV, TDF or TAF) tablet QD orally as per approved package insert.
- Total: Total of all reporting groups
Arm/Group | Virologically Suppressed HBeAg-negative Participants From Parent Study ABI-H0731-201 | Virologically Suppressed HBeAg-positive Participants From Parent Study ABI-H0731-201 | HBeAg Positive Participants From Parent Study ABI-H0731-202 | Total
Number analyzed (Participants) | 26 | 43 | 23 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (7.8) | 45 (11.7) | 36 (13.0) | 44 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of Participants
  Participants
    Female | 10 | 15 | 15 | 40
    Male | 16 | 28 | 8 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 20 | 38 | 22 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 3 | 1 | 1 | 5
  White | 2 | 2 | 0 | 4
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Number of Participants in each location.
  Participants
    New Zealand | 0 | 1 | 1 | 2
    Canada | 0 | 8 | 3 | 11
    Hong Kong | 0 | 1 | 3 | 4
    United States | 26 | 33 | 14 | 73
    United Kingdom | 0 | 0 | 2 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m 2] | 24.38 (2.922) | 23.97 (3.583) | 23.47 (3.984) | 23.96 (3.496)

OUTCOME MEASURES:

1. Primary Outcome: Sustained Viral Response (SVR) at 24 Weeks Off Treatment
Description: To evaluate the potential for combination therapy with ABI-H0731+ NrtI to increase SVR rates in subjects who have chronic hepatitis B (CHB). To evaluate the proportion of subjects who meet the definition of SVR at 24 weeks off treatment, the SVR rate and corresponding 95% confidence interval will be presented for the overall population while on combination therapy.
  SVR is defined as sustained viral response with HBV DNA , LOQ (20 IU/mL) through off-treatment Week 24.
Time Frame: Completing from week 52 until week 76
Population: Participants who met the protocol-specific treatment action criteria to discontinue treatment with ABI-H0731 and NrtI after completing 52 weeks of treatment were analyzed for sustained viral repones at 24 weeks off treatment. (i.e., Completing from week 52 (treatment discharge) until week 76 (24 weeks off treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Virologically-suppressed HBeAg Negative Participants From Parent Study ABI-H0731-201: All participants were treated with ABI-H0731 and NrtI for 52 weeks. Participants without virologic assessment at week 52 were evaluated at the next study visit.
- Virologically-suppressed HBeAg Positive Participants From Parent Study ABI-H0731-201: Participants were treated with ABI-H0731 and NrtI for 52 weeks. Participants without virologic assessment at week 52 were evaluated at the next study visit.
- Treatment-naïve Subjects With HBeAg Positive cHBV: Treatment-naïve subjects with Hepatitis B "e" antigen (HBeAG) positive status with chronic hepatitis B virus (cHBV) from Study ABI-H0731-202 (Parent Study 202)
Arm/Group | Virologically-suppressed HBeAg Negative Participants From Parent Study ABI-H0731-201 | Virologically-suppressed HBeAg Positive Participants From Parent Study ABI-H0731-201 | Treatment-naïve Subjects With HBeAg Positive cHBV
Number analyzed (Participants) | 23 | 18 | 0
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Subjects With Adverse Events
Description: Incidence of treatment emergent adverse events (AEs)
Time Frame: Up to Week 148
Population: Safety population included all who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Virologically-suppressed HBeAg Negative Participants From Parent Study ABI-H0731-201 | Virologically-suppressed HBeAg Positive Participants From Parent Study ABI-H0731-201 | Treatment-naïve Subjects With HBeAg Positive cHBV
Number analyzed (Participants) | 26 | 43 | 23
Participants
  Number of subjects with AEs | 16 | 26 | 12
  Number of subjects with discontinuation due to an AE | 1 | 0 | 2
  Number of subjects with significant abnormal ECGs | 0 | 1 | 0

3. Secondary Outcome: Number of Subjects With Abnormal Alanine Aminotransferase (ALT) at Baseline Who Have Normal ALT at End of Treatment (EOT) and End of Study (EOS)
Description: To measure the number and proportion of subjects with abnormal ALT at baseline who have normal ALT at end of treatment (EOT) and end of study (EOS)
  To measure the number and proportion of subjects regardless of levels of ALT at baseline at EOT and EOS
Time Frame: EOT: up to Week 52 or 148; EOS: up to 3 years off treatment
Population: Number/proportion of subjects with normal alanine aminotransferase (ALT) at end of treatment (EOT) and end of study (EOS)
Measure: Count of Participants; unit: Participants
Arm/Group | Virologically-suppressed HBeAg Negative Participants From Parent Study ABI-H0731-201 | Virologically-suppressed HBeAg Positive Participants From Parent Study ABI-H0731-201 | Treatment-naïve Subjects With HBeAg Positive cHBV
Number analyzed (Participants) | 2 | 2 | 7
Participants
  Numbers with normal ALT levels at EOT | 2 | 0 | 5
  Number with normal ALT levels at EOS | 1 | 0 | 5

4. Secondary Outcome: Number of Subjects With Suppression/Loss of Viral HBeAg Antigen/DNA on Combination Treatment Whose Viral Antigens Rebound Off Therapy
Description: Incidence of subjects with suppression/loss of viral Hepatitis B "e" antigen (HBeAg) antigen/DNA on combination treatment whose viral antigens rebound off therapy
Time Frame: upto Week 148
Population: The proportion of subjects with hepatitis B virus (HBV) DNA target not detected (TND).
  Treatment-naïve Subjects With HBeAg Positive cHBV was not collected. No entry has been made in the column.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment-naïve Subjects With HBeAg Positive cHBV: Treatment-naïve subjects with Hepatitis B "e" Ag antigen (HBeAG) positive status with chronic hepatitis B virus (cHBV) from study ABI-H- (Parent Study 202)
Arm/Group | Virologically-suppressed HBeAg Negative Participants From Parent Study ABI-H0731-201 | Virologically-suppressed HBeAg Positive Participants From Parent Study ABI-H0731-201 | Treatment-naïve Subjects With HBeAg Positive cHBV
Number analyzed (Participants) | 25 | 4 | 0
Participants | 4 | 4 |

5. Secondary Outcome: Number of Subjects With Suppression/Loss of Viral Core-related Antigen/DNA on Combination Treatment Whose Viral Antigens Rebound Off Therapy
Description: Incidence of subjects with suppression/loss of viral core-related antigen (HBcrAg) or DNA on combination treatment whose viral antigens rebound off treatment
Time Frame: Up to Week 148
Population: Subjects from the parent study 201 with positive or negative Hepatitis B "e" antigen (HBeAg)
  Treatment-naïve Subjects With HBeAg Positive cHBV was not collected. No entry has been made in the column.
Measure: Count of Participants; unit: Participants
Arm/Group | Virologically-suppressed HBeAg Negative Participants From Parent Study ABI-H0731-201 | Virologically-suppressed HBeAg Positive Participants From Parent Study ABI-H0731-201 | Treatment-naïve Subjects With HBeAG Positive cHBV
Number analyzed (Participants) | 11 | 0 | 0
Participants | 7 | 0 |

ADVERSE EVENTS:
Time Frame: Up to Week 148
Description: Clinical and laboratory adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version (v) 21.0. System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be provided in the AE dataset. AEs are graded by the Investigator as Grade 1, 2, 3, or 4 according to the toxicity criteria specified in the protocol.
Arm/Group | Virologically Suppressed HBeAg-negative Participants From Parent Study ABI-H0731-201 | Virologically Suppressed HBeAg-positive Participants From Parent Study ABI-H0731-201 | HBeAg Positive Participants From Parent Study ABI-H0731-202
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/43 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/43 | 1/23
Other Adverse Events (participants affected / at risk) | 5/26 | 12/43 | 4/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Virologically Suppressed HBeAg-negative Participants From Parent Study ABI-H0731-201 (N=26) | Virologically Suppressed HBeAg-positive Participants From Parent Study ABI-H0731-201 (N=43) | HBeAg Positive Participants From Parent Study ABI-H0731-202 (N=23)
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Virologically Suppressed HBeAg-negative Participants From Parent Study ABI-H0731-201 (N=26) | Virologically Suppressed HBeAg-positive Participants From Parent Study ABI-H0731-201 (N=43) | HBeAg Positive Participants From Parent Study ABI-H0731-202 (N=23)
upper respiratory tract infection (Infections and infestations) | 3 | 6 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3 | 2
fatique (General disorders) | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT03780543/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT03780543/SAP_001.pdf